CLINICAL TRIAL: NCT05481359
Title: A Post Market, Global Registry to Evaluate the Identification of Atrial Fibrillation Sources Using Electrographic Flow (EGF™) Mapping System to Guide Ablation Therapy in Patients With Atrial Fibrillation in Real-world Setting.
Brief Title: AF-FLOW Registry to Evaluate Electrographic Flow Mapping in Patients Undergoing Ablation for Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Ablacon, Inc. (Industry)
Collaborators: Cortex (Industry)
Responsible Party: Sponsor
Organization: Cortex (Industry)
Other Study IDs: CP-003
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation, Persistent; Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases
Keywords: Electrographic Flow Mapping; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Electrographic Flow™ guided ablation therapy: In addition to standard pulmonary vein isolation (PVI) or PVI touch-up, subjects receive targeted radiofrequency source ablation guided by EGF mapping.
  Interventions: Device: Electrographic Flow™ (EGF) mapping and ablation

INTERVENTIONS:
Device: Electrographic Flow™ (EGF) mapping and ablation — Electrographic Flow™ (EGF) mapping enables the full spatiotemporal reconstruction of organized atrial electrical wavefront propagation to identify active sources or origins of excitation that may trigger atrial fibrillation (AF).
  EGF mapping involves 1 minute recordings of unipolar electrograms from a basket catheter, which are then processed with the EGF algorithm (Ablamap® Software). Several basket catheter positions are acquired in standard positions in both the left and right atria. EGF-identified sources with activity levels exceeding the recommended threshold are deemed significant and are targeted for ablation. The success of the ablation is confirmed through an EGF remap, where elimination of the source is defined as reduction of EGF source activity below the threshold.
  Other Names: Ablamap®; OptiMap™

SUMMARY:
This post-market global registry will evaluate the ability of Electrographic Flow (EGF™) mapping to identify atrial fibrillation (AF) sources and guide ablation therapy in patients with atrial fibrillation in real-world setting.

DETAILED DESCRIPTION:
The AF-FLOW Registry is a prospective, multi-center global post-market registry that will obtain clinical data in order to characterize the performance of Electrographic Flow (EGF™) mapping with Ablamap® Software for its intended use in a real-world setting. Specifically, we will evaluate the ability of EGF mapping to identify sources of atrial fibrillation (AF) and guide ablation therapy in patients with atrial fibrillation. This registry will enroll up to 100 subjects. Subjects that present with AF and meet inclusion/exclusion criteria will be eligible for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Suitable candidate for intra-cardiac mapping and ablation of arrhythmias.
2. Above eighteen (18) years of age or of legal age to give informed consent specific to state and national law.
3. Subjects with a history of documented symptomatic atrial fibrillation.

Exclusion Criteria:

1. Subjects who are not candidates for cardiac ablation procedures.
2. Pregnant or nursing.
3. Presence of anatomic or comorbid conditions, or other medical, social or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or comply with follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from the investigators' general patient population with a history of atrial fibrillation that meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Nilsson, MD, Principal Investigator — Piedmont Athens Hospital
Locations (5):
- United States (3):
  - Piedmont Healthcare, Athens, Georgia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Mount Sinai Hospital, New York, New York
- Erasmus MC, Rotterdam, South Holland, Netherlands
- Medicover Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson KR, Anerao A, Kong MH, Derejko P, Szili-Torok T, Goyal S, Turagam M, Verma A, Castellano S. Electrographic Flow Mapping Provides Prognosis for AF Ablation Outcomes Across Two Independent Prospective Patient Cohorts. J Clin Med. 2025 Jan 22;14(3):693. doi: 10.3390/jcm14030693. PMID 39941362
- [Result] Nilsson KR, Castellano S, Kong MH, Derejko P, Szili-Torok T, Goyal SK, Wijchers S, Turagam M, Reddy VY, Verma A; other members of the AF-FLOW Global Registry Study Group. AF-FLOW Global Registry Confirms Validity of Electrographic Flow Mapping as a Phenotyping Tool for Atrial Fibrillation. J Cardiovasc Electrophysiol. 2025 Mar;36(3):589-599. doi: 10.1111/jce.16568. Epub 2025 Jan 16. PMID 39817626
- [Derived] Kutinsky I, Nilsson KR, Mrlik M, Kong MH, Mehta N, Castellano S. Electrographic flow (EGF) mapping reveals sex-based differences in EGF patterns with women concentrated in phenotypes that benefit from EGF-guided ablation. J Interv Card Electrophysiol. 2026 Jan 7. doi: 10.1007/s10840-025-02184-8. Online ahead of print. PMID 41498861

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrographic Flow™ Guided Ablation Therapy: In addition to standard pulmonary vein isolation (PVI) or PVI touch-up, subjects received targeted radiofrequency source ablation guided by Electrographic Flow™ (EGF) mapping.
Period: Overall Study
Arm/Group | Electrographic Flow™ Guided Ablation Therapy
Started | 25
Subjects With at Least One EGF-identified Source Detected (Subjects with one or more Electrographic Flow™ (EGF) identified source(s) ≥ 26% source activity) | 16
Received EGF-guided Ablation (Subjects who received Electrographic Flow™ (EGF) guided ablation of one or more EGF-identified sources with an activity above threshold) | 13
Did Not Receive EGF-guided Ablation (Subjects who did not receive Electrographic Flow™ (EGF) guided ablation, which included: * Subjects not inducible in AF after pulmonary vein isolation, preventing EGF mapping * Subjects with no EGF-identified sources above threshold on EGF mapping * Subjects where the physician elected not to ablate an EGF-identified source above threshold) | 12
Completed (Completed with 12M Follow-Up) | 21
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Electrographic Flow™ Guided Ablation Therapy: In addition to standard pulmonary vein isolation (PVI) or PVI touch-up, subjects receive targeted radiofrequency source ablation guided by Electrographic Flow™ (EGF) mapping.
Arm/Group | Electrographic Flow™ Guided Ablation Therapy
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 6
  United States | 9
  Poland | 10
Body Mass Index, Continuous [Mean (Standard Deviation); unit: kg/m2] | 27.9 (3.9)
CHA2DS2VASc score, Categorical [Mean (Standard Deviation); unit: units on a scale [scale range: 0-9]] — Tool to describe risk of ischemic stroke in patients with AF. To help guide the decision to treat patients with anticoagulants. Calculated by adding the number of risk factors: Congestive Heart Failure, Hypertension, Age≥75, Diabetes, Stroke/TIA, Vascular Disease, Age 65-74 years and Female Sex. Each risk factor adds a point to the risk score, except for Age ≥ 75 years & Stroke/TIA, which both add 2 points. Score of 0 represents a patient having no additional risk factors. The ESC guidelines considers a score of 1 to be moderate risk and a score ≥ 2 to be high risk. Range: 0 (low) - 9 (high)
  units on a scale [scale range: 0-9] | 2.7 (1.9)
Left Atrial Diameter [Median (Inter-Quartile Range); unit: cm] | 4.4 [3.8 to 4.8]
Left Atrial Volume Index [Median (Inter-Quartile Range); unit: mL/m2] | 40 [29 to 52]
Left Ventricular Ejection Fraction, Continuous [Median (Inter-Quartile Range); unit: %] | 55 [55 to 60]
Paroxysmal AF [Count of Participants; unit: Participants] | 9
Persistent Atrial Fibrillation [Count of Participants; unit: Participants] | 14
Long-standing persistent AF [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Procedure Success
Description: Acute Procedure Success is defined as targeting and successful elimination of significant sources of electrographic flow (EGF) through radiofrequency ablation. EGF-identified sources are significant when their leading source activity is ≥ 26%. Successful elimination is defined as reduction of the source activity of the leading source to <26% upon post-ablation remapping using EGF mapping.
Time Frame: During the procedure
Population: Subjects treated optimally per protocol
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With EGF Identified Sources: Subjects in whom the physician elected to target Electrographic Flow™ (EGF)-identified sources > 26% using RF ablation.
Arm/Group | Subjects With EGF Identified Sources
Number analyzed (Participants) | 13
Participants | 13

2. Secondary Outcome: Number of Participants With 12-month Freedom From AF Recurrence
Description: This measure represents the number of subjects with freedom from documented episodes of atrial fibrillation (AF) recurrence lasting longer than 30 seconds from the 90-day post-procedure blanking period through 12 months of follow-up.
  Only subjects with completed 12 month follow-up are included in this analysis.
Time Frame: 90 day - 12 months
Population: The analysis population for the secondary outcome consisted of two groups:
  Group 1: Subjects who received EGF-guided ablation
  Group 2: Subjects who did not receive EGF-guided ablation, which included:
  * Subjects not inducible in AF after pulmonary vein isolation, preventing EGF mapping
  * Subjects with no EGF-identified sources above threshold (≥26%) on EGF mapping
  * Subjects where the physician elected not to ablate an EGF-identified source above threshold
Measure: Count of Participants; unit: Participants
Groups:
- Subjects That Received EGF-guided Ablation: Subjects who received Electrographic Flow™ (EGF) guided ablation of one or more EGF-identified sources with an activity above threshold
- Subjects That Did Not Receive EGF-guided Ablation: Subjects who did not receive Electrographic Flow™ (EGF) guided ablation, which included:
  * Subjects not inducible in AF after pulmonary vein isolation, preventing EGF mapping
  * Subjects with no EGF-identified sources above threshold on EGF mapping
  * Subjects where the physician elected not to ablate an EGF-identified source above threshold
Arm/Group | Subjects That Received EGF-guided Ablation | Subjects That Did Not Receive EGF-guided Ablation
Number analyzed (Participants) | 11 | 10
Participants | 8 | 6

ADVERSE EVENTS:
Time Frame: From Index Procedure to 12 Month Follow Up
Arm/Group | Subjects That Received EGF-guided Ablation | Subjects That Did Not Receive EGF-guided Ablation
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/12
Other Adverse Events (participants affected / at risk) | 0/13 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects That Received EGF-guided Ablation (N=13) | Subjects That Did Not Receive EGF-guided Ablation (N=12)
Hemorrhage of iliac vein with retroperitoneal hematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects That Received EGF-guided Ablation (N=13) | Subjects That Did Not Receive EGF-guided Ablation (N=12)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
In this real-world registry, the decision to target EGF-identified sources was left to physician discretion. Consequently, numerous EGF-identified sources exceeding the threshold were not ablated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT05481359/Prot_SAP_000.pdf